CLINICAL TRIAL: NCT05997615
Title: A Phase 1, First-in-Human Study of the Safety, Pharmacokinetics, and Preliminary Efficacy of VIR-5500 (AMX-500) in Participants With Prostate Cancer
Brief Title: Safety, Pharmacokinetics, and Preliminary Efficacy of VIR-5500 (AMX-500) in Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vir Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VIR-5500-V101; U1111-1287-6968 (Registry Identifier: ICTRP); 2023-503495-24 (Registry Identifier: CTIS); AMX-500 (Other: Vir Biotechnology, Inc.)
Record Dates: First submitted 2023-07-24; First posted 2023-08-18 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Hormone-refractory Prostate Cancer
Keywords: Prostate Cancer; Castration Resistant Prostatic Cancer; Low-Volume Oligometastatic Hormone Sensitive Prostate Cancer (HSPC); High-Risk Biochemical Recurrent Prostate Cancer; Metastatic Castration-resistant Prostate Cancer (mCRPC)
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Neoplasms, Castration-Resistant | interventions — enzalutamide; darolutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: VIR-5500 Monotherapy Dose Escalation (Experimental): VIR-5500 will be administered as a monotherapy in patients with mCRPC over a 21-day cycle
  Interventions: Drug: VIR-5500
- Part 2: VIR-5500 Monotherapy Dose Expansion (Experimental): VIR-5500 will be administered as a monotherapy in patients with mCRPC over a 21-day cycle
  Interventions: Drug: VIR-5500
- Part 3a: VIR-5500 in combination with an ARSI for Dose Escalation (Experimental)
  Interventions: Combination Product: Enzalutamide; Combination Product: Darolutamide
- Part 4a: VIR-5500 in combination with an ARSI for Dose Expansion (Experimental)
  Interventions: Combination Product: Enzalutamide; Combination Product: Darolutamide

INTERVENTIONS:
Drug: VIR-5500 — Pharmaceutical form: Solution for infusion Route of administration: Intravenous (IV) infusion
  Arms: Part 1: VIR-5500 Monotherapy Dose Escalation; Part 2: VIR-5500 Monotherapy Dose Expansion
Combination Product: Enzalutamide — Oral administration
  Arms: Part 3a: VIR-5500 in combination with an ARSI for Dose Escalation; Part 4a: VIR-5500 in combination with an ARSI for Dose Expansion
Combination Product: Darolutamide — Oral administration
  Arms: Part 3a: VIR-5500 in combination with an ARSI for Dose Escalation; Part 4a: VIR-5500 in combination with an ARSI for Dose Expansion

SUMMARY:
The study will be conducted in 4 parts and will commence with dose escalation of VIR-5500 as a monotherapy (Part 1), followed by combination escalation (Part 3a), monotherapy dose expansion (Part 2) and combination dose expansion (Part 4a).

* Part 1 (Monotherapy Dose Escalation): Single-agent VIR-5500 dose escalation
* Part 2 (Monotherapy Dose Expansion): Single-agent VIR-5500 dose expansion
* Part 3 (Combination Dose Escalation): VIR-5500 plus another therapeutic agent dose escalation

  o Part 3a (Combination Dose Escalation): VIR-5500 in combination with an androgen receptor signaling inhibitor (ARSI) (enzalutamide or darolutamide)
* Part 4 (Combination Dose Expansion): VIR-5500 plus another therapeutic agent dose expansion o Part 4a (Combination Dose Expansion): VIR-5500 in combination with an ARSI (enzalutamide or darolutamide)

DETAILED DESCRIPTION:
Duration of the study up to approximately 48 months.

ELIGIBILITY:
Inclusion Criteria:

Applicable to Parts 1 and 2

* Have metastatic disease, defined by ≥ 1 metastatic lesion that is present on baseline computed tomography (CT), magnetic resonance imaging (MRI), or bone scan imaging
* Have documented progressive mCRPC based on ≥ 1 of the criteria (per PCWG3)
* Have been treated with ≥ 1 second-generation androgen-signaling inhibitor, including abiraterone, apalutamide, darolutamide, and/or enzalutamide
* Have been treated with ≥ 1 prior taxane regimens (e.g., docetaxel, cabazitaxel)
* Are deemed unsuitable for standard of care

Applicable to Part 2 Cohort 1

• Must have received standard-of-care radioligand-based therapies, including PSMA-targeted radiopharmaceutical therapy, such as 177Lu-PSMA-617

Applicable to Part 3a and Part 4a

* Have metastatic CRPC, defined by ≥ 1 metastatic lesion that is present on baseline CT, MRI, or bone scan imaging that has documented progressive disease (PD) based on ≥ 1 of the following criteria (per PCWG3)
* Have metastatic HSPC, defined by at least 1 and no more than 5 metastatic lesions with no visceral involvement that are present on baseline CT, MRI, or bone scan imaging
* Have biochemical recurrent prostate cancer

Exclusion Criteria:

* Presence of dominant histopathological features representative of sarcomatoid, spindle cell, or neuroendocrine small cell components
* Has acute or chronic infections
* Has a concomitant medical or inflammatory condition that may increase the risk of toxicity to VIR-5500, per the Investigator
* Has lesions in proximity of vital organs
* Has known active CNS metastases and/or carcinomatous meningitis The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 390 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2027-09-29 (Estimated); Study Completion 2027-09-29 (Estimated)

PRIMARY OUTCOMES:
Part 1 and 3a: Number of participants with treatment-emergent Adverse Events (AEs) | from the Cycle 1(each cycle is 21 days), Day 1 up to approximately 48 months
  Incidence and severity of AEs according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)
Part 1 and 3a: Incidence of Dose Limiting Toxicities (DLTs) | from the Cycle 1(each cycle is 21 days), Day 1 up to Day 21
  Incidence and nature of DLTs according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)
Part 2 and 4a: Prostate-Specific Antigen (PSA) response rate | from the Cycle 1(each cycle is 21 days), Day 1 up to approximately 48 months
Part 2 and 4a: Objective Response Rate (ORR) | from the Cycle 1(each cycle is 21 days), Day 1 up to approximately 48 months

SECONDARY OUTCOMES:
Part 2 and 4a: Number of participants with Adverse Events (AEs) | from the Cycle 1(each cycle is 21 days), Day 1 up to approximately 48 months
Part 1 and 3a: PSA response rate | from the Cycle 1(each cycle is 21 days), Day 1 up to approximately 48 months
Part 1 and 3a: Objective Response Rate (ORR) | from the Cycle 1(each cycle is 21 days), Day 1 up to approximately 48 months
All parts: Duration of response (DoR) | from the Cycle 1(each cycle is 21 days), Day 1 up to approximately 48 months
All parts: Progression Free Survival PFS | from the Cycle 1(each cycle is 21 days), Day 1 up to approximately 48 months
All parts: Assessment of PK parameters: Cmax | from the Cycle 1(each cycle is 21 days), Day 1 up to approximately 48 months
All parts: Assessment of PK parameters: AUC | from the Cycle 1(each cycle is 21 days), Day 1 up to approximately 48 months
All parts: Assessment of PK parameters: Tmax | from the Cycle 1(each cycle is 21 days), Day 1 up to approximately 48 months
All parts: Incidence of baseline anti-drug antibodies (ADAs) to VIR-5500 | from the Cycle 1(each cycle is 21 days), Day 1 up to approximately 48 months
All parts: Incidence of treatment emergent anti-drug antibodies (ADAs) to VIR-5500 | from the Cycle 1(each cycle is 21 days), Day 1 up to approximately 48 months

CONTACTS AND LOCATIONS:
Locations (8):
- Australia (2):
  - Investigational Site Number: 100, Melbourne
  - Investigational Site Number: 101, Sydney
- Spain (5):
  - Investigational Site Number: 251, Barcelona
  - Investigational Site Number: 250, Barcelona
  - Investigational Site Number: 254, Madrid
  - Investigational Site Number: 252, Madrid
  - Investigational Site Number: 253, Pamplona
- Investigational Site Number: 300, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants.